CLINICAL TRIAL: NCT02048098
Title: A Comparison Between Vaginal Misoprostol vs. Buccal Misoprostol For Second Trimester Termination of Pregnancy
Brief Title: Misoprostol for Second Trimester Termination of Pregnancy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Ragıp Atakan Al, Associate Professor, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: atauni9
Record Dates: First submitted 2014-01-24; First posted 2014-01-29 (Estimated); Last update posted 2015-01-16 (Estimated); Status verified 2015-01

CONDITIONS: Abortion, Induced
Keywords: misoprostol; Labor, Induced; Pregnancy Trimester, Second; Abortion, Induced
MeSH Terms: conditions — Neoplasm Metastasis | interventions — Misoprostol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Buccal misoprostol (Active Comparator): 400 µg buccal misoprostol per 3 hours
  Interventions: Drug: Buccal misoprostol
- vaginal misoprostol (Active Comparator): 400 µg vaginal misoprostol per 3 hours
  Interventions: Drug: Vaginal misoprostol

INTERVENTIONS:
Drug: Vaginal misoprostol — 400 µg vaginal misoprostol per 3 hours up to 6 doses. The treatment will be withold if the patient has strong uterine contractions. If abortion had not occured in 24 hour after the start of the study a second course of 400 µg vaginal misoprostol per 3 hours up to 6 doses will be administered. If abortion had not occured in 48 hour after the start of the study it will be considered treatment failure and patient will be offered another induction/delivery method or to continue protocol.
  Other Names: Cytotec
  Arms: vaginal misoprostol
Drug: Buccal misoprostol — 400 µg buccal misoprostol per 3 hours up to 6 doses. The treatment will be withold if the patient has strong uterine contractions. If abortion had not occured in 24 hour after the start of the study a second course of 400 µg buccal misoprostol per 3 hours up to 6 doses will be administered. If abortion had not occured in 48 hour after the start of the study it will be considered treatment failure and patient will be offered another induction/delivery method or to continue protocol.
  Other Names: Cytotec
  Arms: Buccal misoprostol

SUMMARY:
The purpose of this study is to compare the efficacy of 400 µg vaginal misoprostol per 3 hours to 400 µg buccal misoprostol per 3 hours in second trimester termination of viable pregnancy

ELIGIBILITY:
Inclusion Criteria:

* gestational age between 12-24 weeks
* live fetus
* singleton pregnancy
* Bishop score <5
* no uterine contraction

Exclusion Criteria:

* prostaglandin allergy
* a scar in uterus
* uterine abnormality
* premature rupture of membranes

Ages: 16 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 130 (Actual)
Dates: Start 2014-01; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Induction to fetal expulsion interval | 15 minutes after fetus delivered
  Time elapsed between administration of the first misoprostol dose until expulsion of the fetus

SECONDARY OUTCOMES:
Delivery within 24 hours | 24 hour
Delivery within 48 hours | 48 hours
Use of additional interventions | One week
  the patients who did not delivered within 48 hours will considered as failed induction and will be offered another method of induction/delivery or to continue same protocol.
Expected pain before induction and perceived (actual) pain after abortion completed | within 1 hour after randomisation and after 12 hour after complete abortion/placenta removed
  Expected and perceived pain will be measured by VAS
Rate of complete abortion | 12 hour after fetus and placenta removed

OTHER OUTCOMES:
total misoprostol dose | 48 hours
difference in hematocrit measured at entry of the study and after delivery/abortion | at recruitment and 24 hour after abortion
maternal complications | one weeks
  includes, but not limited blood, transfusions, laparatomy, nausea, vomiting, fever, genital tract injury

CONTACTS AND LOCATIONS:
Overall Officials: Ragıp A AL, MD, Principal Investigator — Ataturk University Faculty of Medicine; Ömer E Yapça, MD, Study Chair — Ataturk University Faculty of Medicine
Locations (1):
- Ataturk Universitesi Araştırma Hastanesi, Erzurum, Turkey (Türkiye)

REFERENCES:
- [Derived] Al RA, Yapca OE. Vaginal Misoprostol Compared With Buccal Misoprostol for Termination of Second-Trimester Pregnancy: A Randomized Controlled Trial. Obstet Gynecol. 2015 Sep;126(3):593-598. doi: 10.1097/AOG.0000000000000946. PMID 26181087